CLINICAL TRIAL: NCT02689596
Title: Intranasal Oxytocin and Resting State fMRI in Healthy Volunteers
Brief Title: Oxytocin and Resting State fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Monika Eckstein, Senior Investigator, University Hospital Heidelberg
Purpose: Basic Science
Other Study IDs: OT-REST14
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
MeSH Terms: interventions — Oxytocin

ARMS (2):
- OT (Active Comparator): Oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: OT
Other: Placebo
  Arms: Placebo

SUMMARY:
The goal of the study is to investigate the effects of intranasal oxytocin (OT) or placebo to resting state brain activity in healthy males.

DETAILED DESCRIPTION:
Although several fMRI studies investigated the neural correlates of OT administration, only few have focused on the underlying modulatory effects of OT on baseline brain function. While functional MRI examines the neural activity during a certain task, it might be especially interesting to assess the main effect of OT on the basic activity of the human brain in rest. This resting state activity becomes typically evident in the default mode network (DMN), compromising midline structures such as medial frontal cortex, cingulate and precuneus, as well as specific resting state networks .

In fact, a recent study succeeded in demonstrating a modulatory influence of OT. Recent studies were able to show an increased functional connectivity at rest of amygdala to the medial prefrontal cortex (PFC) in a small sample of 15 subjects.

However, distinct subregions of the amygdala seem to be involved in different OT effects. To goal of the present study is to decipher the modulatory effects of OT to subregions of the amygdala in a larger sample using improved anatomical mapping of the seed regions and relate these alterations to individual traits of healthy volunteers. We expected to add evidence to the increase of amygdala - PFC connectivity under OT as well as detailed anatomical mapping of this networks.

ELIGIBILITY:
Inclusion Criteria:

* Health

Exclusion Criteria:

* Chronic physical or mental illness, regular smoking or alcohol consumption and medication intake

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2014-10; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Resting state brain activity using fMRI | 30min

SECONDARY OUTCOMES:
Subject personality using questionnaires | 30min